CLINICAL TRIAL: NCT03424733
Title: A Trial of Prednisone and Acetaminophen Versus Acetaminophen Alone in Minimizing Flu-like Symptoms From Pegylated Interferon Beta-1a
Brief Title: Evaluating the Use of Prednisone to Decrease Pegylated Interferon Beta-1a Side Effects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holy Name Medical Center, Inc. (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Mary Ann Picone, MD, Neurologist, Holy Name Medical Center, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: US-PEG-16-10990
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
Keywords: demyelination; relapse rate; Pegylated interferon beta-1a; side effects; flu-like symptoms; injection site reactions; prednisone
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases; Injection Site Reaction | interventions — peginterferon beta-1a; Prednisone; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients in both arms first take Tylenol and then take Tylenol in combination with Prednisone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Current Plegridy Users (Active Comparator): Members in this group have been previously titrated and are currently taking the pegylated interferon beta-1 (Plegridy) injection once every two weeks. These patients will complete a total of six study injections of Plegridy (125 micrograms) totaling a 12 week study duration. Subjects must take two 325mg tablets of Tylenol 1 hour prior to each study injection, and one 20mg Prednisone tablet 4-5 hours prior to injections two through six only.
  Interventions: Drug: Plegridy; Drug: Prednisone; Drug: Tylenol Pill
- New Plegridy Users (Experimental): Members in this group have never taken the pegylated interferon beta-1a (Plegridy) injection, and so they must first by titrated by injecting with a 63 and 94 microgram Plegridy dose. Titrations, along with full dose injections (125 micrograms) occur every two weeks. Patients must take two 325mg tablets of Tylenol prior to each titration injection. The third study dosage involves subjects taking the full 125 microgram Plegridy dosage with two 325mg Tylenol tablets prior to injection. The final five study injections (four through eight) require patients to take two 325mg Tylenol tablets 1 hour prior to injection, and one 20mg Prednisone tablet 4-5 hours prior to injection.
  Interventions: Drug: Plegridy; Drug: Prednisone; Drug: Tylenol Pill

INTERVENTIONS:
Drug: Plegridy — Self injection into area of high adipose content. Injections include 63 and 94 microgram titration doses, and the full 125 microgram dose
  Other Names: Pegylated Interferon beta-1a
Drug: Prednisone — Take one 20 milligram prednisone tablet four to five hours prior to injections two through six of the full 125 microgram Plegridy dose.
Drug: Tylenol Pill — Take two 325 milligram Tylenol tablets 1 hour prior to each Plegridy injection, irregardless of dosage.
  Other Names: Acetaminophen

SUMMARY:
Some of the most common side effects of the multiple sclerosis drug Plegridy (pegylated interferon beta-1a) include flu-like symptoms and injection site reactions. Physicians often advise patients to take Tylenol or aspirin prior to injection, but in this study the investigators evaluated whether using a low dose of oral steroid in combination with Tylenol reduced flu-like symptoms and injection site reactions.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic neurological disease characterized by demyelination of the brain and spine. Currently, there are several treatments designed to decrease the frequency of attacks and delay disease progression. One of these treatments, interferon beta, has shown the potential to decrease relapse rates by approximately 30%, but because the body quickly clears these proteins, patients require more frequent dosing. Another interferon therapy called pegylated interferon beta-1a (Plegridy) was released and it was shown to last longer in the body than interferon beta-1a. This is why Plegridy can be take by an injection into tissue under the skin once every 14 days. However, some of the most common side effects of interferon beta therapy include flu-like symptoms and injection skin reactions, which can often cause patients to want to stop treatment. Clinical practitioners often advise patients to take acetaminophen (Tylenol) or aspirin before the injection in order to prevent the onset or decrease the severity of flu-like symptoms. A previous study with patients taking interferon beta-1a showed that taking a low dose oral steroid (prednisone) in addiction to a medication like Tylenol reduced flu-like symptoms compared to just taking Tylenol by itself. Because Plegridy lasts longer in the body and has more convenient dosing for patients, researchers in this study decided to investigate whether taking prednisone in addition to acetaminophen before the injection would help decrease or prevent the occurrence of flu-like symptoms and injection site reactions in patients taking the therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed any form of MS (relapsing remitting, primary progressive, secondary progressive), any EDSS (expanded stability status scale) score

Exclusion Criteria:

* prior allergic reaction to interferon products, congestive heart failure, elevated liver enzymes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Flu-like symptoms | 12 to 16 weeks
  Reduced flu-like symptoms from Plegridy injections due to taking both Tylenol and Prednisone prior to treatment. Flu-like symptoms are measured every 6 hours for 48 hours after injection by patients self reporting their muscle aches, temperature, chills, and fatigue on a Holy Name administered Flu-like symptom questionnaire.

SECONDARY OUTCOMES:
Injection site reactions | 12 to 16 weeks
  Reduced injection site reactions from Plegridy injections due to taking both Tylenol and Prednisone prior to injection. Injection site reactions are reported to a clinical research assistant approximately one week after injection. If present, patients must record their injection site reactions using a Holy Name administered tape measurer in centimeters, as well as descriptive characteristics of the injection (location on body, swelling, redness, itching, and pain). The clinical research assistant records all of the data on an injection site reaction form.

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rio J, Nos C, Marzo ME, Tintore M, Montalban X. Low-dose steroids reduce flu-like symptoms at the initiation of IFNbeta-1b in relapsing-remitting MS. Neurology. 1998 Jun;50(6):1910-2. doi: 10.1212/wnl.50.6.1910. PMID 9633761
- [Result] Brandes DW, Bigley K, Hornstein W, Cohen H, Au W, Shubin R. Alleviating flu-like symptoms with dose titration and analgesics in MS patients on intramuscular interferon beta-1a therapy: a pilot study. Curr Med Res Opin. 2007 Jul;23(7):1667-72. doi: 10.1185/030079907x210741. PMID 17588298
- [Result] Rio J, Nos C, Bonaventura I, Arroyo R, Genis D, Sureda B, Ara JR, Brieva L, Martin J, Saiz A, Sanchez Lopez F, Prieto JM, Roquer J, Dorado JF, Montalban X. Corticosteroids, ibuprofen, and acetaminophen for IFNbeta-1a flu symptoms in MS: a randomized trial. Neurology. 2004 Aug 10;63(3):525-8. doi: 10.1212/01.wnl.0000133206.44931.25. PMID 15304586